CLINICAL TRIAL: NCT05436314
Title: The Effectiveness of Manual Lymphatic Drainage in Fibromyalgia Syndrome
Brief Title: Manual Lymphatic Drainage in Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Gamze Kurt, Ph.D., Kutahya Health Sciences University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: MLDfibro
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; pain; manual lymphatic drainage
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual Lymphatic Drainage Group (Experimental): Manual Lymphatic Drainage (MLD) in addition to medical treatment is applied to participants in this group.
  Interventions: Other: Manual Lymphatic Drainage; Drug: Medical treatment
- Sham Group (Sham Comparator): Sham Manual Lymphatic Drainage (MLD) in addition to medical treatment is applied to participants in this group.
  Interventions: Drug: Medical treatment; Other: Sham Manual Lymphatic Drainage

INTERVENTIONS:
Other: Manual Lymphatic Drainage — Manual Lymphatic Drainage (MLD) is applied towards the flow direction of lymph vessels with special hand movements. MLD is made with very light, completely painless and rhythmic translational movements of the skin. MLD, by expert and trained physiotherapists (G.K, H.K) in this field. It will be applied with the techniques defined by Dr. Vodder. MLD ( to the neck region, abdominal region, axillary and inguinal lymph nodes) will be applied by following the lymphatic pathways specific to the anterior and posterior trunk, respectively. The treatment session will take approximately 45 minutes. It will be applied 5 days a week during 3 weeks.
  Arms: Manual Lymphatic Drainage Group
Drug: Medical treatment — The patients in control group continued taking their regular gabapentin and pregabalin-derivative drug therapy at the same dosage and duration specified by their physicians.
Other: Sham Manual Lymphatic Drainage — Sham MLD will be administered by MLD-trained physiotherapists (G.K, H.K) with a protocol that is far from techniques that reveal the physiological effects of MLD. Sham application consists of applications that do not follow the lymphatic pathways from distal to proximal to the trunk, neck, and abdominal region, and superficial breathing. The session will take approximately 45 minutes.
  Arms: Sham Group

SUMMARY:
There are limited studies on the use of Manual Lymphatic Drainage (MLD) in fibromyalgia syndrome. Considering the possible mechanisms of action of MLD and the pathophysiology of fibromyalgia, more studies are needed to fully determine the effect of MLD on this syndrome. The aim of this study was to investigate the effectiveness of manual lymphatic drainage on symptom severity, pain intensity, pressure pain threshold and anxiety about pain in fibromyalgia syndrome.

DETAILED DESCRIPTION:
Fibromyalgia Syndrome (FMS) is a syndrome of unknown cause, characterized by numerous symptoms such as chronic widespread pain, fatigue, insomnia, joint stiffness, depression, concentration and memory problems, myofascial pain and tender points. The prevalence of FMS in the general population is 2%, and it is a common syndrome. There are studies showing that there is dysfunction in the connective tissue or fascia in FMS that triggers peripheral nociceptor stimulation. Any change in fascial tissue motility can cause an imbalance between body fluids leading to tissue hardening and accumulation of toxins. By stimulating the lymph vessels, metabolic waste products can be eliminated, excess fluid can be reduced, blockages can be removed and the immunological system can be regulated. Pharmacological and non-pharmacological methods are used in the treatment of FMS. Exercise, manual therapy techniques, cognitive behavioral treatments, patient education and other physiotherapy modalities are the non-pharmacological methods that are frequently used. Manual lymphatic drainage (MLD) was developed in 1965 by Dr. It is a manual therapy technique that consists of slow, rhythmic, superficial and repetitive movements defined by Vodder. Many effects that MLD can reveal locally and systemically are discussed. MLD; It stimulates the lymphatic and parasympathetic system, reduces pain, helps regulate the immune system, clears blockages, eliminates metabolic wastes and toxins in the body, and reduces excess fluid. There are limited studies on the use of MLD in fibromyalgia syndrome. Considering the possible mechanisms of action of MLD and the pathophysiology of fibromyalgia, more studies are needed to fully determine the effect of MLD on this syndrome. The aim of this study was to investigate the effectiveness of manual lymphatic drainage on symptom severity, pain intensity, pressure pain threshold and anxiety about pain in fibromyalgia syndrome.

ELIGIBILITY:
Inclusion Criteria:

* have fibromyalgia as defined by the criteria of the 2016 ACR
* have Turkish as their native language
* between 18 and 65 years of age

Exclusion Criteria:

* Having cognitive impairment
* Receiving routine physiotherapy and/or manual therapy, alternative/complementary therapies
* Illiterate people
* Diagnosed with endocrine, neuromuscular, infectious and inflammatory diseases
* Diagnosed severe mental and psychological disorders
* Having malignancy
* Pregnant or people who breastfeed

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire (FIQ) | 5 minutes
  The FIQ is an assessment and evaluation instrument developed to measure fibromyalgia (FM) patient status, progress and outcomes.
Pressure pain thresholds (PPT) | 10 minutes
  Pressure pain thresholds in following three points, 7th cervical vertebra,6th thoracal vertebra and 3th lumbal vertebra were measured using a analog pressure algometer (Baseline, USA).
Visual Analogue Scale | 1 minutes
  A 0-100mm Visual Analogue Scale (VAS) will be used to assess pain intensity. The VAS is a scale on a straight line with a value of "0" indicating "no pain intensity" and a value of "100" indicating "severe pain". Participants will be asked to mark the pain they feel on this line.

SECONDARY OUTCOMES:
Concerns About Pain | 5 minutes
  Participants' concerns about painwill be evaluated with the "Washington University Pain-Related Worries Scale (UWCAP-TR)", which was recently developed as a pain self-efficacy measure based on modern scale development approaches and adapted into Turkish by Saraçoğlu et al. UWCAP-TR consists of 8 questions and 2 parts. While the first part of the scale evaluates concerns about pain, the second part evaluates the individual's self-confidence in the face of pain. The scores of each section are collected and evaluated separately. Scoring of the scale is done with a 5-point Likert type scale. The first part is scored between 6-30, the second part is scored between 2-10. High scores on the UWCAP-TR indicate increased anxiety about pain and low confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze KURT, Ph.D., Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University Evliya Celebi Hospital, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No